CLINICAL TRIAL: NCT02220426
Title: Phase 1 Study: Detection of Brown Adipose Tissue in Normal Volunteers Using a 3 Tesla (3T) Magnetic Resonance Imaging System and Hyperpolarized (HP) Xenon Gas
Brief Title: Hyperpolarized Xenon-129 Magnetic Resonance Imaging and Spectroscopy of Brown Fat: Healthy Adult Volunteer Pilot Study
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: North Carolina Translational and Clinical Sciences Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 14-1211
Record Dates: First submitted 2014-08-15; First posted 2014-08-19 (Estimated); Results first posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-09

CONDITIONS: Obesity
Keywords: Brown adipose tissue; Hyperpolarized xenon gas MRI
MeSH Terms: conditions — Obesity | interventions — Xenon

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Xenon inhalation (Other): Inhalation up to 5 doses of 750ml of hyperpolarized 129Xe gas
  Interventions: Drug: Xenon

INTERVENTIONS:
Drug: Xenon — Inhalation of hyperpolarized xenon gas
  Other Names: Hyperpolarized xenon gas

SUMMARY:
The primary goal of this study is to evaluate the feasibility of detecting Brown Adipose Tissue (BAT) in healthy subjects by using hyperpolarized xenon gas MRI.

In this pilot study, MRI of BAT of healthy adult volunteers will be performed at 3 Tesla to assess image quality using a prototype surface coil and pulse sequence following inhalation of hyperpolarized 129Xe (xenon) gas at thermoneutrality and under mild cold condition.

The investigators are testing the abilities of xenon MRI to see brown adipose tissue and detect its thermogenic activity.

DETAILED DESCRIPTION:
In the fight against obesity, brown adipose tissue (BAT) is considered to be the newest target. The hypothesis is that this tissue is partially responsible for the imbalance between energy intake and energy expenditure that keeps lean people lean and obese people obese.

As the detection of this tissue in adult humans is difficult, this study aim to evaluate the use of hyperpolarized xenon gas MRI for the detection of this tissue.

Hyperpolarized xenon gas MRI is currently used for lung ventilation studies. For this study subjects will undergo an MRI scan for which they will also inhaled hyperpolarized xenon. Scans will be done before and during stimulation of thermogenic activity by cold exposure, while MR images and spectra will be acquired from the supraclavicular area. We expect that the inhaled gas will diffuse into blood and eventually reach BAT in a manner proportional to the metabolic activity of this tissue.

Objectives of this studies are:

* To detect BAT volume using hyperpolarized xenon MRI
* To detect BAT thermogenic activity by hyperpolarized xenon Nuclear Magnetic Resonance (NMR) spectroscopy

ELIGIBILITY:
Inclusion Criteria:

* Ability to give informed consent
* Willing to participate in this study
* Male or female ≥ 18 years of age at the time of the interview.
* Subject has no diagnosed pulmonary condition
* Subject has not smoked in the previous 5 years
* Smoking history, if any, is less than or equal to 5 pack-years
* Written informed consent (and assent when applicable) obtained from subject or subject's
* legal representative and ability for subject to comply with the requirements of the study
* Healthy subject that may or may not have undergone an fluorodeoxyglucose -Positron Emission Tomography (PET) scan

Exclusion Criteria:

* Any contraindication to MRI (presence of any non-removable metal implant, stents, pacemaker, clips, staples, or piercings, etc. )
* Subject does not fit in the magnet
* Pregnancy or breast feeding
* Severe claustrophobia
* Subject is less than 18 years old
* MRI is contraindicated based on responses to MRI screening questionnaire
* Subject is pregnant or lactating
* Respiratory illness of a bacterial or viral etiology within 15 days of MRI
* Subject has received an investigational medicinal product (not including 129Xe) within 30 days of MRI
* Subject has any form of known cardiovascular disease
* Subject cannot hold their breath for 15 seconds
* Subject deemed unlikely to be able to comply with instructions during imaging
* Subject is taking beta blockers
* Subject underwent an fluorodeoxyglucose-PET examination less than one week before the HP xenon MRI scan

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2016-07-01 (Actual); Study Completion 2016-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rosa Tamara Branca, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Biomedical Research Imaging Center, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Branca RT, He T, Zhang L, Floyd CS, Freeman M, White C, Burant A. Detection of brown adipose tissue and thermogenic activity in mice by hyperpolarized xenon MRI. Proc Natl Acad Sci U S A. 2014 Dec 16;111(50):18001-6. doi: 10.1073/pnas.1403697111. Epub 2014 Dec 1. PMID 25453088

RESULTS

PARTICIPANT FLOW:
Groups:
- Xenon Inhalation: Inhalation of up to 5 doses of 750ml of hyperpolarized 129Xe gas
  Xenon: Inhalation of hyperpolarized xenon gas
Period: Overall Study
Arm/Group | Xenon Inhalation
Started | 17
Signed Informed Consent | 17
Received Xenon Inhalation | 13
Completed | 13
Not Completed | 4

BASELINE CHARACTERISTICS:
Arm/Group | Xenon Inhalation
Number analyzed (Participants) | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.6 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 13
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 11
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 13

OUTCOME MEASURES:

1. Primary Outcome: Brow Adipose Tissue Surface Area
Description: For each subject, the brown adipose tissue (BAT) surface area is derived from 2D MR images acquired without slice selection, obtained before and during cold exposure. Each image consists of Nx × Ny pixels, each having an in-plane pixel area (Apixel, in millimeters squared) calculated as: Apixel=(FOVx/Nx)×(FOVy/Ny), where FOVx and FOXy are the field-of-view dimensions in millimeters in the x and y directions, respectively. BAT-positive pixels are defined as those whose signal intensity increases by more than 5% during cold stimulation relative to baseline.
  The total BAT surface area (ABAT, in millimeters squared) is then computed as:
  ABAT=NBAT×Apixel where NBAT is the number of BAT-positive pixels for each subject.
  This approach yields the total in-plane area of activated BAT within the 2D field of view for each subject. The value obtained for all subjects was then averaged.
Time Frame: Day 1
Population: No imaging data were collected for 9 participants because the Xenon signal did not reach the needed threshold required for imaging.
Measure: Mean (Standard Deviation); unit: millimiters squared
Units Other Than Participants: 2-D images
Groups:
- Xenon Inhalation: Inhalation of 5 doses of 750ml of hyperpolarized 129Xe gas
  Xenon: Inhalation of hyperpolarized xenon gas
Arm/Group | Xenon Inhalation
Number analyzed (Participants) | 4
Number analyzed (2-D images) | 7
millimiters squared | 3541 (2474)

2. Secondary Outcome: Change in BAT Temperature
Description: Change in BAT temperature (in degree Celsius) will be estimated from xenon nuclear magnetic resonance (NMR) spectra acquired at thermoneutrality and during cold exposure. Both proton (1H) and xenon (129Xe) spectra are required to perform the temperature calculation.
Time Frame: Day 1
Population: Temperature measurements were not performed because the xenon and proton spectra were acquired with different magnet settings, which prevented alignment of the signals required for calculation.
Arm/Group | Xenon Inhalation
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Within two minutes after xenon inhalation and continuing through and ending at one hour after the last xenon inhalation, a total of up to 1 hour in total.
Arm/Group | Xenon Inhalation
All-Cause Mortality (participants affected / at risk) | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 12/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Xenon Inhalation (N=13)
Restlessness (Nervous system disorders) | 1 (1)
Numbness (Nervous system disorders) | 8 (8)
Euphoria (Psychiatric disorders) | 2 (2)
Tingling (Nervous system disorders) | 8 (8)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Lightheadedness (Nervous system disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 5 (5)
Device site discomfort (Injury, poisoning and procedural complications) | 5 (5) — Discomfort on finger from pulse oximeter
Somnolence (sleepiness) (Nervous system disorders) | 2 (2)
Chest discomfort (twinge following inhalation) (Cardiac disorders) | 1 (1)
Increase in blood pressure prior inhalation (Vascular disorders) | 1 (1)
Back pain from lying in scanner (Musculoskeletal and connective tissue disorders) | 1 (1)
Dizziness (Nervous system disorders) | 6 (6)

LIMITATIONS AND CAVEATS:
This pilot study was conducted to optimize the magnetic resonance protocol for detecting hyperpolarized xenon gas dissolved in brown adipose tissue (BAT). As no prior human data were available, early participants were studied to refine the protocol and identify possible issues with the magnetic resonance imaging and spectroscopy protocol.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-10-09): https://cdn.clinicaltrials.gov/large-docs/26/NCT02220426/Prot_SAP_000.pdf